CLINICAL TRIAL: NCT06284798
Title: A First Human Dose Study Investigating Safety, Tolerability, and Pharmacokinetics of Subcutaneous Single Ascending Doses of NNC0650-0013 in Healthy Male Participants
Brief Title: A Research Study of a New Medicine (NNC0650-0013) in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9650-5027; 2023-506134-79 (Other: European Medical Agency (EMA)); U1111-1291-7535 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NNC0650-0013: Subcutaneous dose (Experimental): Participants will receive NNC0650-0013 subcutaneously in an ascending dose manner.
  Interventions: Drug: NNC0650-0013 A
- Placebo (Placebo Comparator): Participants will receive matching placebo to NNC0650-0013 subcutaneously.
  Interventions: Drug: Placebo
- NNC0650-0013: Intravenous dose (Experimental): Participants will receive NNC0650-0013 in an ascending dose manner intravenously.
  Interventions: Drug: NNC0650-0013 A

INTERVENTIONS:
Drug: NNC0650-0013 A — NNC0650-0013 will be administered subcutaneously or intravenously.
  Arms: NNC0650-0013: Intravenous dose; NNC0650-0013: Subcutaneous dose
Drug: Placebo — Subcutaneous administration.
  Arms: Placebo

SUMMARY:
This study is testing a new study medicine which may be used to treat people with type 2 diabetes. NNC0650-0013 is a new medicine, which cannot be prescribed by doctors. The purpose of the study is to see if the new study medicine is safe, and how it works in participants body. Participants will get a single dose of the study medicine either as injection(s) under the skin or into a vein. The injection will be given by the study staff. If participants are chosen to get the study medicine as injections under the skin, participants will either get NNC0650-0013 or placebo (a "dummy medicine" without any active ingredients). Which treatment participants get is decided by chance. Participants will be required to fast overnight 3 times during the study. The study will last between 11 and 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index between 24.0 and 29.9 kilogram per meter square (kg/m^2) (both inclusive) at screening.
* Considered to be otherwise healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, unwillingness or inability, which, in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) greater than or equal to 6.5 percent (48 millimoles per mole (mmol/mol)) at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
S.C. Cohort: Number of treatment emergent adverse events (TEAEs) | From time of dosing (day 1) until completion of the follow-up visit (day 75)
  Measured as number of events.

SECONDARY OUTCOMES:
S.C. Cohort: AUC0-∞,0188,SD: Area under the NNC0519-0188 plasma concentration time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow up visit (day 75)
  Measured as hours nanomoles per liter (h*nmol/L).
S.C. Cohort: Cmax,0188,SD: Maximum plasma concentration of NNC0519-0188 after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as nanomoles per liter (nmol/L).
S.C. Cohort: AUC0-∞,0013,SD: Area under the NNC0650-0013 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as h*nmol/L.
S.C. Cohort: Cmax,0013,SD: Maximum observed plasma concentration of NNC0650-0013 after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as nanomoles per liter (nmol/L).
S.C. Cohort: AUC0-∞,0031,SD: Area under the NNC0650-0031plasma concentration time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as h*nmol/L.
S.C. Cohort: Cmax,0031,SD: Maximum observed plasma concentration of NNC0650-0031 after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as nanomoles per liter (nmol/L).
I.V. Cohort: AUC0-∞,0188,SD: Area under the NNC0519-0188 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as h*nmol/L.
I.V. Cohort: AUC0-∞,0013,SD: Area under the NNC0650-0013 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as h*nmol/L.
I.V. Cohort: AUC0-∞,0031,SD: Area under the NNC0650-0031 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) until completion of the follow-up visit (day 75)
  Measured as h*nmol/L.
S.C. and I.V. Cohort: AUC0-∞,0013,SD/dose: Area under the NNC0650-0013 plasma concentration-time curve from time 0 to infinity after a single dose divided by the dose administered | From pre-dose (day1) until completion of the follow-up visit (day 75)
  Measured as hours nanomoles per milligram (h*nmol/mg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency' (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com